CLINICAL TRIAL: NCT05371665
Title: A Native Path to Courage: Feasibility Study of a Culturally Adapted Emotional-Behavioral Prevention Program for American Indian Children
Brief Title: Feasibility of a Culturally Adapted Emotional-Behavioral Prevention Program for American Indian Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Brandon Scott, Associate Professor, Montana State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: bscott; 5P20GM104417 (NIH)
Record Dates: First submitted 2022-04-12; First posted 2022-05-12 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Anxiety Disorder; Depressive Disorder
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Culturally Adapted Cognitive-Behavioral Prevention and Early Intervention (PEI) Program (Experimental): All youth received the culturally adapted prevention and early intervention program from trained providers in the school setting.
  Interventions: Behavioral: Culturally Adapted Cognitive-Behavioral Prevention and Early Intervention (PEI) Program

INTERVENTIONS:
Behavioral: Culturally Adapted Cognitive-Behavioral Prevention and Early Intervention (PEI) Program — The prevention and early intervention is originally an indicated cognitive-behavioral program for 8-13-year-old youth with higher anxiety. Our CAB adapted it as a universal prevention and early intervention for all American Indian youth in the tribal community. It was delivered across six weeks with 20-30 min weekly sessions. Youth engaged in games and role-play reducing anxiety and stress in mildly challenging situations to provide in-vivo exposure. Session 1 involved introductions, relaxation training, and discussing emotions. Session 2 taught youth about worries and how to handle them. Session 3 focused on having conversations with others. Session 4 taught youth how to be assertive (CAB identified this as an area of adaption in initial meetings). Session 5 taught youth how to face their fears. Session 6 was a review session. Parents and teachers were sent notes of what youth learned in each session and asked to encourage youth to practice their learned skills.

SUMMARY:
American Indians (AI) are at greater risk for anxiety and depression early in life. This is concerning given the potential negative effects of these conditions across the lifespan (substance use, suicide). Available culturally adapted prevention and early interventions (PEIs) for anxiety and depression in AI youth are limited. Thus, there is a critical need for the development and evaluation of a culturally consonant, brief PEI for anxiety and depression in AI youth. The investigators' goal is to provide the community with a potentially successful PEI to mitigate AI youth's anxiety and depression that integrates culture and traditions for delivery in schools. The Specific Aims of the proposed research were to 1) culturally adapt a PEI program for AI youth living on a Northern Plains tribal reservation (chosen by the Cultural Advisory Board; CAB), 2) evaluate the feasibility and acceptability of the culturally-adapted program with AI youth living on the reservation, and 3) estimate effect size changes in anxiety and depressive symptoms of the culturally adapted program with the AI youth. The investigators built upon the investigators' strong community relationships and CBPR methods to achieve these aims. The investigators partnered with the CAB to culturally adapt the PEI program for AI youth in year 1 and 2 using a CBPR framework, including AI youth and parents. In year 2, the investigators trained an AI school counselor from the tribal community and a white school counselor from the two tribal serving schools on the reservation to implement the adapted PEI program. We pilot tested the 6-week program (one 20-30 minute session per week) with 28 AI 3rd-6th graders in two schools serving youth from the reservation in year 3. The investigators will partner with the tribal community to further refine and tailor the adapted PEI program using the results of this study. Moreover, further testing of the refined program's efficacy and sustainability will be conducted using a larger sample and randomized, two-group design.

DETAILED DESCRIPTION:
American Indians (AI) are at greater risk for anxiety and depression early in life. This is concerning given the potential negative effects of these conditions across the lifespan (substance use, suicide). Available culturally adapted prevention and early interventions (PEIs) for anxiety and depression in AI youth are limited. Thus, there is a critical need for the development and evaluation of a culturally appropriate, brief PEI for anxiety and depression in AI youth. These were the three main goals of this study: 1) Partner with a Northern Plains tribal community to culturally adapt the PEI program for AI youth living on the reservation. 2) evaluate whether they were able to successfully provide the program to AI youth in two tribal schools and whether youth would accept/enjoy the program, and 3) test whether there were changes in anxiety and depressive symptoms, as well as resilience, among the AI youth from pre- to post-intervention. The investigators partnered with the tribal community, including AI youth and parents, to culturally adapt the PEI program in years 1 and 2. In year 3, the investigators trained an AI school counselor from the tribal community and a white school counselor to provide the adapted PEI program in the two tribal-serving schools. Twenty-eight AI 3rd-6th graders (8-12 years-old) participated in the program. The investigators will continue to partner with the tribal community to further refine and tailor the culturally adapted program using the results from this study. Moreover, further testing of the refined program's efficacy and sustainability will be conducted using a larger sample and control group.

This study built upon a community-based participatory research partnership with a Northern Plains tribal community to culturally adapt a brief and evidence-based prevention and early intervention (PEI) program addressing anxiety and depression in American Indian (AI) 8-12-year-olds. The investigators evaluated how feasible it would be for AI providers from the tribal community to deliver the adapted intervention to AI youth attending two schools serving the tribe. The investigators also tested the hypotheses that AI youth will find the program acceptable and enjoyable, and it will reduce anxiety and depressive symptoms from pre- to post-intervention.

The investigators used an iterative adaptation process within a CBPR framework to culturally adapt the evidence-based PEI program. It involved collaborating with the Cultural Advisory Board (CAB) and conducting adult work groups and youth focus groups with keys community stakeholders, including AI youth and parents, to determine cultural adaptations and adapt the program. The investigators first collaborated with the CAB in reviewing prior literature on anxiety and depression, as well as the non-adapted PEI program. The CAB developed an initial conceptual model of what factors may cause or put AI youth at risk for anxiety and depression. In addition the model included what outcomes were expected from a prevention and early intervention program targeting these causal or risk factors. Next, they used AI cultural and tribal specific knowledge to modify the model integrate the understanding and meaning of anxiety and depression and behavioral determinants and outcomes from their tribal and cultural perspective. This involved adding, removing, or modifying/replacing certain parts of the initial model to better align with the tribe's worldview of mental health and healing. Moreover, the CAB identified cultural or tribal behavioral determinants (e.g., cultural identity) of anxiety and depression not described in the literature and add them to the model.

Next, the investigators recruited 20 community stakeholders (Elders, parents/legal guardians, and mental health specialists who serve the community) and 14 AI 8-12 year-olds to review the non-adapted intervention and suggest cultural adaptions and improvements to the content, strategies, and materials. Focus groups were audio recorded. Youth also completed a pre-adaptation usability survey (they reviewed only 3 of the 6 program modules) of the non-adapted PEI program that assessed acceptability, enjoyableness, and cultural appropriateness.

The investigators analyzed focus and work group discussions to identify common themes and group suggestions together. The CAB used this information and integrate with their own suggestions to: 1) modify a conceptual framework of anxiety and depression prevention and early intervention in AI youth, and 2) determine the cultural adaptations that are most warranted given possible logistical barriers (e.g., time/funding). Identified themes were reviewed and validated with the CAB and Project Manager. The CAB worked with the research team to culturally adapt the intervention and identified two school counselors (i.e., an American Indian tribal member and a white non-tribal member) to provide it in the schools.

The two school counselors provided the program to 28 AI youth in the 3rd to 6th grade (8-12 years-old) in the two schools that serve the tribal community. The adapted intervention was delivered once a week for six weeks and each session lasted 20-30 minutes. Youth completed a post-adaption usability survey at the end of each session to assess acceptability and likeability of the adapted program. The investigators also collected survey data on the primary and secondary measures 1 week before the intervention (pre) and 1 week following the intervention (post). Survey data was collected electronically using a tablet or computer and included: youth demographics, the primary outcomes of youth anxiety and depressive symptoms (from youth and teachers), and secondary outcomes that include youth resilience, youth's beliefs whether they can control their anxiety symptoms, and youth's use of rumination when sad. The CAB worked with the research team using the conceptual model in the adaptation process to decide on the addition, removal, or further revision of the assessments. The youth who completed the intervention and were present for session 6 participated in a post-intervention focus (3-4 youth per group) to further discuss their experiences with adapted intervention and suggest improvements. The focus groups were audio recorded. The two intervention providers also recorded youth attendance and provided additional information about following the program guidelines and steps as trained, what material was covered or not covered, and their judgements on implementing the program.

ELIGIBILITY:
Inclusion Criteria:

• 8-12 year-old youth who attends either tribe-serving school and resides on the reservation with their parent/legal guardian.

Exclusion Criteria:

• Does not meet inclusion criteria.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montana State University, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No
The study data is owned by the tribal community and we would need their permission to share data with other researchers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Elders/parents/teachers/mental health professionals were not considered enrolled in the study. Only youth were enrolled in the study.
Groups:
- Culturally Adapted Prevention and Early Intervention Program: All youth received the culturally adapted prevention and early intervention from trained providers in the school setting.
Period: Overall Study
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Started | 28
Completed | 26
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: One participant did not complete the baseline or outcome measures. However, the participant did attend sessions 2 and 3 before not returning for sessions 4 to 6. The participant was counted as dropping out of the program. Another participant completed the baseline and outcomes measures, but did not attend sessions 3 to 6 and was counted as dropping out of the program.
  Baseline data was not collected for adults. Teachers only reported baseline data on youth.
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: One participant did not complete the baseline or outcome measures. However, the participant did attend sessions 2 and 3 before not returning for sessions 4 to 6. The participant was counted as dropping out of the program. Another participant completed the baseline and outcomes measures, but did not attend sessions 3 to 6 and was counted as dropping out of the program.
  Years | 10.19 (1.10)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant did not complete the baseline or outcome measures. However, the participant did attend sessions 2 and 3 before not returning for sessions 4 to 6. The participant was counted as dropping out of the program. Another participant completed the baseline and outcomes measures, but did not attend sessions 3 to 6 and was counted as dropping out of the program.
  Participants
    Female | 14
    Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant did not complete the baseline or outcome measures. However, the participant did attend sessions 2 and 3 before not returning for sessions 4 to 6. The participant was counted as dropping out of the program. Another participant completed the baseline and outcomes measures, but did not attend sessions 3 to 6 and was counted as dropping out of the program.
  Participants
    American Indian or Alaska Native | 21
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 4
    Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity measure included a category for "Hispanic." Results reported are for those participants who either reported they were "Hispanic" or another race/ethnicity.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 26
    Unknown or Not Reported | 0
Youth-reported Anxiety Disorder Symptoms [Mean (Standard Deviation); unit: mean score on scale] — The Revised Child Anxiety and Depression Scale - Short Version Child Report (RCADS-25-S) is a 25-item instrument used to assess DSM-IV anxiety disorders symptoms (15 items) and depressive disorder symptoms (10 items). Youth rated how often each anxiety and depressive disorder symptom is true of them on a rating scale consisting of: 0 (Never), 1 (Sometimes), 2 (Often), and 3 (Always). Mean scores range from 0 to 3 with higher mean scores indicating greater frequency of youths' anxiety disorder symptoms. Population: Two youth did not attend 4 or more sessions and were not included in outcome measure analysis.
  mean score on scale | .95 (.44)
Youth-reported Depressive Disorder Symptoms [Mean (Standard Deviation); unit: mean score on scale] — The Revised Child Anxiety and Depression Scale - Short Version Child Report (RCADS-25-S) is a 25-item instrument used to assess DSM-IV anxiety disorders symptoms (15 items) and depressive disorder symptoms (10 items). Youth rated how often each anxiety and depressive disorder symptom is true of them on a rating scale consisting of: 0 (Never), 1 (Sometimes), 2 (Often), and 3 (Always). Mean scores range from 0 to 3 with higher mean scores indicating greater frequency of youths' depressive disorder symptoms. Population: Two youth did not attend 4 or more sessions and were not included in outcome measure analysis.
  mean score on scale | 1.08 (.51)
Teacher-reported Anxiety Disorder Symptoms [Mean (Standard Deviation); unit: mean score on scale] — The Revised Child Anxiety and Depression Scale - Short Version Teacher Report is a 25-item instrument used to assess DSM-IV anxiety disorders symptoms (15 items) and depressive disorder symptoms (10 items). Teachers rated how often each anxiety and depressive disorder symptom is true of each youth on a rating scale consisting of: 0 (Never), 1 (Sometimes), 2 (Often), and 3 (Always). Mean scores range from 0 to 3 with higher mean scores indicating greater frequency of youths' anxiety disorder symptoms. Population: Two teachers did not complete the measure at pre-intervention. One teacher did not complete the measure at post-intervention for certain youth. Some teachers did were missing 20% of the required items for the mean scale score to be calculated at either pre- or post-intervention.
  mean score on scale
    number analyzed (Participants) | 11
    (all) | .33 (.25)
Teacher-reported Depressive Disorder Symptoms [Mean (Standard Deviation); unit: mean score on scale] — The Revised Child Anxiety and Depression Scale - Short Version Teacher Report is a 25-item instrument used to assess DSM-IV anxiety disorders symptoms (15 items) and depressive disorder symptoms (10 items). Teachers rated how often each anxiety and depressive disorder symptom is true of each youth on a rating scale consisting of: 0 (Never), 1 (Sometimes), 2 (Often), and 3 (Always). Mean scores range from 0 to 3 with higher mean scores indicating greater frequency of youths' depressive disorder symptoms. Population: Two teachers did not complete the measure at pre-intervention. One teacher did not complete the measure at post-intervention for certain youth. Some teachers did were missing 20% of the required items for the mean scale score to be calculated at either pre- or post-intervention.
  mean score on scale
    number analyzed (Participants) | 16
    (all) | .43 (.32)
Youth-reported Anxiety Control Beliefs [Mean (Standard Deviation); unit: mean score on scale] — The Anxiety Control Questionnaire for Children assesses children's control beliefs over anxiety-related "external" threats (e.g., fear-producing objects, events, and situations) and/or "internal" emotional or bodily reactions (e.g., flushed face). Youth rated how much each statement was true of them on a 5-point Likert-type scale consisting of: 0 (None), 1 (A Little), 2 (Some), 3 (A Lot), or 4 (Very Very Much). Mean scores range from 0 to 4 with higher mean scores indicate greater perceived control over their anxiety symptoms and external anxiety-related events. Population: Two youth did not attend 4 or more sessions and were not included in outcome measure analysis.
  mean score on scale | 2.25 (.93)
Youth-reported Rumination [Mean (Standard Deviation); unit: mean score on scale] — The Child Response Style Questionnaire - Rumination Scale is 13 item rumination subscale of the 26 item measure. Youth rated how often they engage in each strategy when feeling sad (e.g., "When I am sad, I think about how alone I feel.") on a 4-point scale consisting of "Almost Never" (coded 0), "Sometimes" (coded 1), "Often" (coded 2), and "Almost Always" (coded 3). Mean rumination scale scores ranged from 0 to 3 with higher mean scale scores indicating greater rumination. Population: Two youth did not attend 4 or more sessions and were not included in outcome measure analysis.
  mean score on scale | 1.46 (.60)
Youth-reported Personal Skills Resilience [Mean (Standard Deviation); unit: mean score on scale] — The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' personal skills. Population: Two youth did not attend 4 or more sessions and were not included in outcome measure analysis.
  mean score on scale | 1.46 (.29)
Youth-reported Peer Support Resilience [Mean (Standard Deviation); unit: mean score on scale] — The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' peer support. Population: Two youth did not attend 4 or more sessions and were not included in outcome measure analysis.
  mean score on scale | 1.31 (.57)
Youth-reported Social Skills Resilience [Mean (Standard Deviation); unit: mean score on scale] — The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' social skills. Population: Two youth did not attend 4 or more sessions and were not included in outcome measure analysis.
  mean score on scale | 1.62 (.37)
Youth-reported Physical Caregiving Resilience [Mean (Standard Deviation); unit: mean score on scale] — The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' physical caregiving. Population: Two youth did not attend 4 or more sessions and were not included in outcome measure analysis.
  mean score on scale | 1.44 (.50)
Youth-reported Psychological Caregiving Resilience [Mean (Standard Deviation); unit: mean score on scale] — The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' psychological caregiving. Population: Two youth did not attend 4 or more sessions and were not included in outcome measure analysis.
  mean score on scale | 1.56 (.39)
Youth-reported Spiritual Resilience [Mean (Standard Deviation); unit: mean score on scale] — The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' spiritual experiences. Population: Two youth did not attend 4 or more sessions and were not included in outcome measure analysis.
  mean score on scale | 1.54 (.40)
Youth-reported Educational Resilience [Mean (Standard Deviation); unit: mean score on scale] — The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' educational experiences. Population: Two youth did not attend 4 or more sessions and were not included in outcome measure analysis.
  mean score on scale | 1.42 (.39)
Youth-reported Cultural Resilience [Mean (Standard Deviation); unit: mean score on scale] — The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' cultural experiences. Population: Two youth did not attend 4 or more sessions and were not included in outcome measure analysis.
  mean score on scale | 1.38 (.33)
Youth-reported Tribal Specific Resilience [Mean (Standard Deviation); unit: mean score on scale] — The Child and Youth Resilience Measure - Tribal Resilience Scale is a 10-item measure that assesses tribal specific resilience based on exposure or using Native language, exposure or knowing Native/tribal history, and exposure or experiencing tribal or cultural practices. Youth indicated to what extent each statement describes them or their experiences on a three-point scale of 0 ("Not at All"), 1 ("Somewhat") and 2 ("A Lot"). Mean scale scores range from 0 to 2 with higher scores reflecting greater tribal specific resilience as it pertains to youths' tribal and cultural experiences. Population: Two youth did not attend 4 or more sessions and were not included in outcome measure analysis.
  mean score on scale | 1.20 (.34)

OUTCOME MEASURES:

1. Primary Outcome: Post-Intervention Youth-reported Anxiety Disorder Symptoms From Pre- to Post-Intervention
Description: The Revised Child Anxiety and Depression Scale - Short Version Child Report (RCADS-25-S) is a 25-item instrument used to assess DSM-IV anxiety disorders symptoms (15 items) and depressive disorder symptoms (10 items). Youth rated how often each anxiety and depressive disorder symptom is true of them on a rating scale consisting of: 0 (Never), 1 (Sometimes), 2 (Often), and 3 (Always). Mean scores range from 0 to 3 with higher mean scores indicating greater frequency of youths' anxiety disorder symptoms at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
mean score on scale | .94 (.65)

2. Other Pre Specified Outcome: Mean Likability of the Prevention and Early Intervention Modules
Description: Youth completed a usability survey at the end of each intervention 30-minute module (Modules 1, 2, 3, 4, and 5) that measured the likeability of that specific module. Youth rated how much they liked the entire lesson for that module on a three-point scale consisting of 1 ("Did Not Like"), 2 ("Liked") and 3 ("Very Much Liked "). A mean likability score (ranging from 1 to 3) was calculated for each module with higher mean scores indicating greater likeability of that module.
Time Frame: Assessed at Completion of Each 30-minute Module
Population: The number of participants analyzed for each module is different due to certain participants not attending that specific session.
  Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
Score on a scale
  Module 1: number analyzed (Participants) | 23
  Module 1 | 2.43 (.51)
  Module 2: number analyzed (Participants) | 22
  Module 2 | 2.5 (.51)
  Module 3: number analyzed (Participants) | 20
  Module 3 | 2.5 (.51)
  Module 4: number analyzed (Participants) | 21
  Module 4 | 2.6 (.50)
  Module 5: number analyzed (Participants) | 24
  Module 5 | 2.33 (.57)

3. Primary Outcome: Post-Intervention Youth-reported Depressive Disorder Symptoms
Description: The Revised Child Anxiety and Depression Scale - Short Version Child Report (RCADS-25-S) is a 25-item instrument used to assess DSM-IV anxiety disorders symptoms (15 items) and depressive disorder symptoms (10 items). Youth rated how often each anxiety and depressive disorder symptom is true of them on a rating scale consisting of: 0 (Never), 1 (Sometimes), 2 (Often), and 3 (Always). Mean scores range from 0 to 3 with higher mean scores indicating greater frequency of youths' depressive disorder symptoms at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
mean score on scale | 1.03 (.51)

4. Secondary Outcome: Post-Intervention Youth-reported Anxiety Control Beliefs
Description: The Anxiety Control Questionnaire for Children assesses children's control beliefs over anxiety-related "external" threats (e.g., fear-producing objects, events, and situations) and/or "internal" emotional or bodily reactions (e.g., flushed face). Youth rated how much each statement was true of them on a 5-point Likert-type scale consisting of: 0 (None), 1 (A Little), 2 (Some), 3 (A Lot), or 4 (Very Very Much). Mean scores range from 0 to 4 with higher mean scores indicate greater perceived control over their anxiety symptoms and external anxiety-related events at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: One participant was missing more than 20% of items on the ACQ-C measure at post-intervention and thus a mean score could not be a calculating resulting in the mean being based on 25 youth.
  Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 25
mean score on scale | 2.42 (.66)

5. Secondary Outcome: Post-Intervention Youth-reported Rumination
Description: The Child Response Style Questionnaire - Rumination Scale is 13 item rumination subscale of the 26 item measure. Youth rated how often they engage in each strategy when feeling sad (e.g., "When I am sad, I think about how alone I feel.") on a 4-point scale consisting of "Almost Never" (coded 0), "Sometimes" (coded 1), "Often" (coded 2), and "Almost Always" (coded 3). Mean rumination scale scores ranged from 0 to 3 with higher mean scale scores indicating greater rumination at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
mean score on scale | 1.22 (.70)

6. Secondary Outcome: Post-Intervention Youth-reported Personal Skills Resilience
Description: The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' personal skills at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
mean score on scale | 1.35 (.33)

7. Secondary Outcome: Post-Intervention Youth-reported Peer Support Resilience
Description: The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' peer support at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
mean score on scale | 1.50 (.60)

8. Secondary Outcome: Post-Intervention Youth-reported Social Skills Resilience
Description: The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' social skills at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
mean score on scale | 1.52 (.36)

9. Secondary Outcome: Post-Intervention Youth-reported Physical Caregiving Resilience
Description: The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' physical caregiving at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
mean score on scale | 1.44 (.52)

10. Secondary Outcome: Post-Intervention Youth-reported Psychological Caregiving Resilience
Description: The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' psychological caregiving.
Time Frame: Post-Intervention
Population: Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
mean score on scale | 1.58 (.36)

11. Secondary Outcome: Post-Intervention Youth-reported Spiritual Resilience
Description: The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' spiritual experiences at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
mean score on scale | 1.46 (.56)

12. Secondary Outcome: Post-Intervention Youth-reported Educational Resilience
Description: The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' educational experiences at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
mean score on scale | 1.58 (.39)

13. Secondary Outcome: Post-Intervention Youth-reported Cultural Resilience
Description: The Child and Youth Resilience Measure is a 26-item measure that assesses resiliency across a number of domains. Youth indicated to what extent each statement describes them (e.g., "Getting an education is important to me," "I try to finish activities that I start," and "I feel supported by my friends") on a three-point scale of 0 ("No"), 1 ("Sometimes") and 2 ("Yes"). Mean scale scores range from 0 to 2 with higher mean scale scores reflecting greater resilience as it pertains to youths' cultural experiences at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
mean score on scale | 1.38 (.36)

14. Primary Outcome: Post-Intervention Teacher-reported Anxiety Disorder Symptoms
Description: The Revised Child Anxiety and Depression Scale - Short Version Teacher Report is a 25-item instrument used to assess DSM-IV anxiety disorders symptoms (15 items) and depressive disorder symptoms (10 items). Teachers rated how often each anxiety and depressive disorder symptom is true of each youth on a rating scale consisting of: 0 (Never), 1 (Sometimes), 2 (Often), and 3 (Always). Mean scores range from 0 to 3 with higher mean scores indicating greater frequency of youths' anxiety disorder symptoms at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: Teachers only reported on youth outcomes. Although there were 26 youth enrolled in the program, one teacher did not complete the measure at post-intervention for 3 of the youth. In addition, teacher-reported data on five of the youth were missing 20% of the required items for the mean scale score to be calculated at post-intervention. Thus, only 18 youth data was analyzed out of the 26 who were enrolled and analyzed overall.
  Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 18
mean score on scale | .25 (.20)

15. Primary Outcome: Post-Intervention Teacher-reported Depressive Disorder Symptoms
Description: The Revised Child Anxiety and Depression Scale - Short Version Teacher Report is a 25-item instrument used to assess DSM-IV anxiety disorders symptoms (15 items) and depressive disorder symptoms (10 items). Teachers rated how often each anxiety and depressive disorder symptom is true of each youth on a rating scale consisting of: 0 (Never), 1 (Sometimes), 2 (Often), and 3 (Always). Mean scores range from 0 to 3 with higher mean scores indicating greater frequency of youths' depressive disorder symptoms at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: Teachers only reported on youth outcomes. Although there were 26 youth enrolled in the program, one teacher did not complete the measure at post-intervention for 3 of the youth. Thus, only 23 youth data was analyzed out of the 26 who were enrolled and analyzed overall.
  Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 23
mean score on scale | .31 (.26)

16. Other Pre Specified Outcome: Mean Enjoyability of Compass for Courage Modules
Description: Youth completed a usability survey at the end of each intervention 30-minute module (Modules 1, 2, 3, 4, and 5) that measured the enjoyability of that specific module. Youth rated how much fun the entire lesson was for that module on a three-point scale consisting of 1 ("Not Fun"), 2 ("Fun") and 3 ("Very Much Fun"). A mean enjoyability score (ranging from 1 to 3) was calculated for each module with higher mean scores indicating greater enjoyability of that module.
Time Frame: Assessed at Completion of Each 30-minute Module
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
Score on a scale
  Module 1: number analyzed (Participants) | 22
  Module 1 | 2.36 (.58)
  Module 2: number analyzed (Participants) | 22
  Module 2 | 2.36 (.58)
  Module 3: number analyzed (Participants) | 20
  Module 3 | 2.45 (.51)
  Module 4: number analyzed (Participants) | 21
  Module 4 | 2.52 (.51)
  Module 5: number analyzed (Participants) | 24
  Module 5 | 2.38 (.50)

17. Secondary Outcome: Post-Intervention Youth-reported Tribal Specific Resilience
Description: The Child and Youth Resilience Measure - Tribal Resilience Scale is a 10-item measure that assesses tribal specific resilience based on exposure or using Native language, exposure or knowing Native/tribal history, and exposure or experiencing tribal or cultural practices. Youth indicated to what extent each statement describes them or their experiences on a three-point scale of 0 ("Not at All"), 1 ("Somewhat") and 2 ("A Lot"). Mean scale scores range from 0 to 2 with higher scores reflecting greater tribal specific resilience as it pertains to youths' tribal and cultural experiences at post-intervention, 8 weeks post-baseline.
Time Frame: Post-Intervention
Population: Youth are the only participants being assessed.
Measure: Mean (Standard Deviation); unit: mean score on scale
Arm/Group | Culturally Adapted Prevention and Early Intervention Program
Number analyzed (Participants) | 26
mean score on scale | 1.23 (.41)

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Culturally Adapted Cognitive-Behavioral Prevention and Early Intervention (PEI) Program: All youth will receive the culturally adapted COMPASS for Courage from trained providers in the school setting.
  Culturally Adapted Cognitive-Behavioral Prevention and Early Intervention (PEI) Program: COMPASS for Courage is an indicated cognitive-behavioral prevention and early intervention program for 8-13-year-old youth with higher anxiety. Our CAB has decided to adapt it as a universal prevention and early intervention for all American Indian youth in the tribal community. It is delivered across six weeks with 30 min weekly sessions. Youth engage in games and role-play reducing anxiety and stress in mildly challenging situations to provide in-vivo exposure. Session 1 involves introductions, relaxation training, and discussing emotions. Session 2 teaches youth about worries and how to handle them. Session 3 focuses on having conversations with others. Session 4 teaches youth how to be assertive (CAB identified this as an area of adaption in initial meetings). Session 5 teaches youth how to face their fears. Session 6 is a review session. Parents and teachers are sent notes of what youth learned in each session and asked to encourage youth to practice their learned skills.
Arm/Group | Culturally Adapted Cognitive-Behavioral Prevention and Early Intervention (PEI) Program
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT05371665/Prot_SAP_000.pdf